CLINICAL TRIAL: NCT03543072
Title: A Prospective Observational Study About Adjuvant or Neoadjuvant Chemotherapy Related Adverse Effects in Postmenopausal Women With Breast Cancer
Brief Title: A Prospective Observational Study About Adjuvant or Neoadjuvant Chemotherapy Related Adverse Effects in Postmenopausal Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Other Study IDs: SCBCG-022
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diphosphonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposure group: exposed to some factors
  Interventions: Drug: Bisphosphonates
- control group: not exposed to some factors

INTERVENTIONS:
Drug: Bisphosphonates — a class of drugs that prevent the loss of bone density, used to treat osteoporosis and similar diseases
  Groups: exposure group

SUMMARY:
Breast cancer is one of the most common malignant tumor in women. About 69.75% of breast cancer women patients in China are over 45 years old. It is a multicenter prospective observational study. We collect the basic information, medical history, chemotherapy-related adverse reactions, and the results of blood lipid and bone density test before, during and after adjuvant or neoadjuvant chemotherapy. The purpose of the study is to investigate the risk factors for hyperlipidemia, cardiovascular disease, and osteoporosis in postmenopausal breast cancer patients before and after chemotherapy, and to assess the risk of future arteriosclerotic cardiovascular disease and osteoporotic fractures. In addition, the collected information of the subjects are analyzed to provide suggestions for the relevant prevention strategy.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignant tumor in women. About 69.75% of breast cancer women patients in China are over 45 years old. Chemotherapy is one of the important treatments for breast cancer, but it brings a series of adverse effects, especially increasing the risk of hyperlipidemia, cardiovascular disease and osteoporosis in postmenopausal women. It is a multicenter prospective observational study. The postmenopausal breast cancer women patients who are planning adjuvant or neoadjuvant chemotherapy are enrolled in the study after signing the informed consent form and passing the screening. We collect the basic information, medical history, chemotherapy-related adverse reactions, and the results of blood lipid and bone density test before, during and after chemotherapy. The purpose of the study is to investigate the risk factors for hyperlipidemia, cardiovascular disease, and osteoporosis in postmenopausal breast cancer patients before and after chemotherapy, and to assess the risk of future arteriosclerotic cardiovascular disease and osteoporotic fractures in this population.In addition, the collected information of the subjects are analyzed to provide suggestions for the relevant prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form has been signed.
2. Breast cancer patients whose age is ≥ 18 years old and have been diagnosed by histological examination.
3. Postmenopausal women who are defined by any of the following:

   * Previous bilateral oophorectomy;
   * Age ≥ 60 years old;
   * Age <60 years old, menopause at least 12 months, and follicle stimulating hormone [FSH] and estradiol levels in the postmenopausal range.
4. Plan for adjuvant or neoadjuvant chemotherapy.

Exclusion Criteria:

1. Those who have already received adjuvant or neoadjuvant chemotherapy.
2. Those who have chemotherapy contraindications.
3. Those who have any mental condition that prevents the understanding of the contents of this study and can't provide the complete information required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with breast cancer who plan for adjuvant or neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
The rate of osteoporosis | 5 years
  According to the result of bone mineral density

SECONDARY OUTCOMES:
The risk of osteoporotic fracture | 5 years
  Calculate the risk of osteoporotic fracture with the WHO Fracture Risk Assessment Tool (FRAX® ) (http://www.shef.ac.uk/FRAX/)

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided